CLINICAL TRIAL: NCT04499118
Title: A Randomized Phase 2 Trial to Assess the Efficacy of AT in Comparison to TP as Neoadjuvant Chemotherapy in Patients With HER2-negative Early Breast Cancer : Evaluating the Homologous Recombination Deficiency(HRD) Biomarker
Brief Title: AT Versus TP as Neoadjuvant Chemotherapy in Patients With HER2-negative Early Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sichuan Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Luojing, Prof., Sichuan Provincial People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BCHRD201
Record Dates: First submitted 2020-07-28; First posted 2020-08-05 (Actual); Last update posted 2020-08-05 (Actual); Status verified 2020-07

CONDITIONS: HER2-negative Breast Cancer
Keywords: Breast neoplasms; HER2-; Homologous Recombination Deficiency
MeSH Terms: conditions — Breast Neoplasms | interventions — Anthracyclines; Paclitaxel; TP protocol; Platinum

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Arm a(HR+/HER2-,HRD-） (Experimental): Participants receive AT regimen for neoadjuvant therapy
  Interventions: Drug: AT regimen
- Arm b(TNBC, HRD-) (Experimental): Participants receive TP regimen for neoadjuvant therapy
  Interventions: Drug: TP regimen
- Arm c(HER2-,HRD+) (Experimental): Participants receive AT regimen for neoadjuvant therapy
  Interventions: Drug: AT regimen
- Arm d(HER2-, HRD+) (Experimental): Participants receive TP regimen for neoadjuvant therapy
  Interventions: Drug: TP regimen

INTERVENTIONS:
Drug: AT regimen — Doxorubin 60mg/㎡ d1 or Epirubicin 75mg/㎡ d1 Docetaxel 75mg/㎡ d1 1/21d
  Other Names: Anthracycline/Paclitaxel
  Arms: Arm a(HR+/HER2-,HRD-）; Arm c(HER2-,HRD+)
Drug: TP regimen — Albumin paclitaxel 125mg/㎡ d1, 8 Cisplatin 75mg/㎡ d1-3 1/21d✖6 or carboplatin AUC6 d1 1/21d✖6
  Other Names: Paclitaxel/Platinum
  Arms: Arm b(TNBC, HRD-); Arm d(HER2-, HRD+)

SUMMARY:
This is a prospective, randomized and open-label phase II study, evaluating the efficacy and safety of AT vs TP regimen as neoadjuvant treatment for early HER2-negative breast cancer. Participants will undergo/receive HRD testing after enrollment. HRD-positive patients will be randomly assigned in a ratio of 1:1 to receive AT（Doxorubicin or Epirubicin+docetaxel）or TP（Albumin paclitaxel + Cisplatin or Carboplatin）regimen respectively, followed by surgery. HRD-negative patients will be assigned to receive TP（Albumin paclitaxel + Cisplatin or Carboplatin）regimen if TNBC, or AT（Doxorubicin or Epirubicin+docetaxel）rigemen, followed by surgery.

DETAILED DESCRIPTION:
This study intends to adopt Simon's two-stage optimal design. In stage 1, 15 HRD-positive and 15 HRD-negative patients will be recruited to receive AT or TP regimen as neoadjuvant therapy. If more than 5 patients in the HRD-positive group achieve pCR(pathological complete response) , the trial expands to stage 2, otherwise the trial terminates. In stage 2, another 31 HRD- positive and 31 HRD-negative patients will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent for all study specific procedures according to local regulatory requirements prior to beginning specific protocol procedures.
* Age ≥ 18 years.
* Male or female patients
* ECOG performance status ≤1
* Histologically confirmed invasive breast cancer by core needle or incisional biopsy (excisional biopsy is not allowed). Clinical stage T2-3 N0-2 or T1 N1-2 by physical exam or radiologic studies. In case of bilateral cancer, the investigator has to decide prospectively which side will be evaluated for the primary endpoint.
* Centrally confirmed negative HER2-status. Centrally confirmed estrogen and progesterone receptor, and Ki-67 status detected on core biopsy. ER/PR positive is defined as ≥1% stained cells and HER2-positive is defined as IHC 3+ or in-situ hybridisation (ISH) ratio ≥2.0.
* Provide Formalin-fixed, paraffin-embedded (FFPE) breast tissue to take Homologous Recombinant Deficiency test.
* Tumor lesion in the breast with a palpable size of > 2 cm or a sonographical size of >1 cm in maximum diameter. If the tumor is not detectable with sonography mammography assessment can be considered. The lesion has to be measurable in two dimensions, preferably by sonography. In case of inflammatory disease, the extent of inflammation can be used as measurable lesion.
* Normal cardiac function must be confirmed by ECG and cardiac ultrasound (LVEF or shortening fraction) within 3 months prior to randomization. Results must be above the normal limit of the institution.
* Laboratory requirements:

  i. Hematology b) Absolute neutrophil count (ANC) ≥2.0 x 109 / L and c) Platelets ≥100 x 109 / L and d) Hemoglobin ≥10 g/dL (≥ 6.2 mmol/L) Hepatic function e) Total bilirubin ≥1.5x UNL and f) ASAT (SGOT) and ALAT (SGPT) ≥1.5x UNL and g) Alkaline phosphatase ≥2.5x UNL.
* Negative pregnancy test (urine or serum) within 14 days prior to randomization for all women of childbearing potential.
* Patients with a prior history of contra-lateral breast cancer are eligible if they have no evidence of recurrence of their initial primary breast cancer within the last 5 years.
* Individuals with a history of other malignancies are eligible if they have been disease-free for at least 5 years and are deemed by the investigator to be at low risk for recurrence of that malignancy and did not receive prior chemotherapy. Individuals with the following cancers are eligible if diagnosed and treated within the past 5 years: cervical cancer in situ, and basal cell or squamous cell carcinoma of the skin.
* Patients must be available and compliant for central diagnostics, treatment and follow-up.
* Patient must be willing to undergo mandatory research biopsy and blood draw. Prior to biopsy procedures patients must be able to be off medications that could increase the risk of bleeding

Exclusion Criteria:

* Prior chemotherapy for any malignancy within 3 years.
* Any prior treatment for the current breast cancer, including chemotherapy, hormonal therapy, radiation or experimental therapy.
* Ongoing use of any other investigational or study agents.
* Previous malignant disease without being disease-free for less than 5 years (except CIS of the cervix and non-melanomatous skin cancer).
* Renal dysfunction for which exposure to cisplatin would be unsafe or require cisplatin dose modification (i.e., Cre > 1.5 mg/dl or GFR < 60 cc/min).
* Inadequate general condition (not fit for anthracycline-taxane-targeted agents-based chemotherapy).
* Evidence of metastasis before randomization
* Known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS) related diseases, active or symptomatic viral hepatitis or chronic liver disease
* Known history of heart disease, for example: myocardial infarction or symptomatic cardiac ischemia within 24 weeks before screening; congestive heart failure; randomized history of clinically significant ventricular arrhythmias within the previous year; Mobitz II level 2 Or a history of tertiary heart block, hypertension is uncontrolled
* History of significant neurological or psychiatric disorders including psychotic disorders, dementia or seizures that would prohibit the understanding and giving of informed consent.
* Have undergone major surgery within 14 days before entering the study
* Any other reason the investigator considers inappropriate to participate in this clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-08 (Estimated); Primary Completion 2021-08 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Complete pathological response of breast and lymph nodes (ypT0/is ypN0; defined as no microscopic evidence of residual invasive viable tumor cells in all resected specimens of the breast and axilla) | 24 weeks
  1. To compare the pathologic response to neoadjuvant AT regimen in HER2- breast cancer with and without HR-deficiency, defined as a high HRD score or a BRCA mutation
  2. To compare the pathologic response to neoadjuvant TP regimen in HER2- breast cancer with and without HR-deficiency, defined as a high HRD score or a BRCA mutation
  3. To compare the pathologic response to neoadjuvant AT vs TP regimen in HER2- breast cancer with HR-deficiency, defined as a high HRD score or a BRCA mutation

SECONDARY OUTCOMES:
Imaging response | 24 weeks
  To determine the response rates of the breast tumor and axillary nodes based on imaging tests. (sonography, mammography, or MRI) after treatment.
Residual cancer burden in patients with HRD | up to 24 weeks
  RCB in the breast tissue and the lymph node tissue will be performed after the completion of neoadjuvant systemic therapy.
response by pCR in HRD high versus tBRCA | 24 weeks
  To assess the pCR rate in HRD high with vs without tBRCA mutation

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Luojing, Principal Investigator — Sichuan Provincial People's Hospital
Locations (1):
- Department of breast surgery, Sichuan Provincial People's Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tutt A, Tovey H, Cheang MCU, Kernaghan S, Kilburn L, Gazinska P, Owen J, Abraham J, Barrett S, Barrett-Lee P, Brown R, Chan S, Dowsett M, Flanagan JM, Fox L, Grigoriadis A, Gutin A, Harper-Wynne C, Hatton MQ, Hoadley KA, Parikh J, Parker P, Perou CM, Roylance R, Shah V, Shaw A, Smith IE, Timms KM, Wardley AM, Wilson G, Gillett C, Lanchbury JS, Ashworth A, Rahman N, Harries M, Ellis P, Pinder SE, Bliss JM. Carboplatin in BRCA1/2-mutated and triple-negative breast cancer BRCAness subgroups: the TNT Trial. Nat Med. 2018 May;24(5):628-637. doi: 10.1038/s41591-018-0009-7. Epub 2018 Apr 30. PMID 29713086
- See also: Prediction of pathological complete response (pCR) by Homologous Recombination Deficiency (HRD) after carboplatin-containing neoadjuvant chemotherapy in patients with TNBC: Results from GeparSixto. — http://ascopubs.org/doi/abs/10.1200/jco.2015.33.15_suppl.1004
- See also: GeparOLA: paclitaxel+olaparib vs paclitaxel/carboplatin followed by epirubicin/cyclophosphamide in HER2-/HRD+ early breast cancer — http://ascopubs.org/doi/abs/10.1200/JCO.2019.37.15_suppl.506